CLINICAL TRIAL: NCT00967655
Title: A Phase II Study to Evaluate the Efficacy and Safety of Neoadjuvant Radiation in Combination With Capecitabine & Paniumumab With and Without Irinotecan in Patients With Localized Rectal Cancer
Brief Title: Capecitabine, Panitumumab, and Radiation Therapy With or Without Irinotecan Hydrochloride in Treating Patients Undergoing Surgery for Localized Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loma Linda Oncology Medical Group, Inc. (Other)
Responsible Party: Imtiaz A. Malik, Loma Linda Oncology Medical Group, Incorporated
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000652936; LLOMGI-20050743; MALIK 012009
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-09

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Panitumumab; Capecitabine; Irinotecan; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Biological: panitumumab
Drug: capecitabine
Drug: irinotecan hydrochloride
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy, monoclonal antibody therapy, and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying the side effects of giving capecitabine and panitumumab together with radiation therapy with or without irinotecan hydrochloride and to see how well it works in treating patients undergoing surgery for localized rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the pathological tumor response rate in patients with localized rectal cancer treated with neoadjuvant chemoradiotherapy comprising capecitabine, panitumumab, and radiotherapy with or without irinotecan hydrochloride.
* To assess the incidence of grade 3/4 toxicity during neoadjuvant chemoradiotherapy.

Secondary

* To assess the disease-free survival.
* To assess the time to treatment failure.
* To assess the1-year and 2-year survival rates.
* To assess local recurrence, defined as recurrence in pelvis at the site of previous disease.
* To assess the safety and toxicity grade using NCI CTCAE v3.0 criteria.
* To assess the number and percentage of patients who undergo down staging of their disease as determined before initiating neoadjuvant therapy and at the time of surgery.
* To assess the number and percentage of patients where permanent colostomy can be avoided as determined by the surgeon before initiating neoadjuvant therapy and at the time actual surgery is performed.

OUTLINE: This is a multicenter study.

* Phase A: Patients undergo radiotherapy once daily 5 days a week and receive oral capecitabine twice daily 5 days a week for 5½ weeks. Patients also receive panitumumab IV over 1 hour on days 1, 15, and 29 during radiotherapy in the absence of disease progression or unacceptable toxicity.
* Phase B: Patients undergo radiotherapy and receive capecitabine and panitumumab as in Phase A. Patients also receive irinotecan hydrochloride IV on days 1, 8, 22, and 29 in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery 6-8 weeks after completion of chemoradiotherapy,

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the distal rectum (0-9 cm from the dentate line or 3-12 cm from the anal verge)
* T3 or T4 tumor or nodal involvement by endorectal ultrasound or CT scan or MRI

  * Patients with any T status where tumor is close to but not involving the sphincter who otherwise would be candidates for abdominoperineal resection are eligible
* No known homozygotes to UGT1A1* 28
* No distant metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 3 times ULN
* Serum creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 50 mL/min
* Magnesium normal
* Able to tolerate major surgery
* Able and willing to comply with study requirements
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks (males) or 24 weeks (females) after completion of study therapy
* No prior diagnosis of interstitial lung disease
* No prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to fluorouracil
* No other prior or concurrent invasive malignancy unless disease-free for ≥ 5 years
* No lack of physical integrity of the upper gastrointestinal tract, inability to swallow tablets, or malabsorption syndrome
* No concurrent serious infections
* No clinically significant cardiovascular disease within the past year, including any of the following:

  * Myocardial infarction
  * Unstable angina
  * Symptomatic congestive heart failure
  * Symptomatic coronary artery disease
  * Serious uncontrolled cardiac arrhythmia
* No history of any medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase risks associated with study participation or investigational product(s) administration or may interfere with the interpretation of the study results
* No known positivity for HIV, hepatitis C, or acute or chronic active hepatitis B

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for rectal cancer
* No prior anti-EGFr antibody therapy (e.g., cetuximab)
* No prior treatment with small molecule EGFr inhibitors (e.g., gefitinib, erlotinib hydrochloride, or lapatinib ditosylate)
* No prior therapeutic radiotherapy to the pelvis
* More than 28 days since prior major surgery
* More than 14 days since prior minor surgery
* At least 30 days since prior investigational agent or therapy
* At least 4 weeks since prior and no concurrent sorivudine or brivudine
* No concurrent chronic immunosuppressive agents (e.g., methotrexate or cyclosporine)
* No concurrent cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate
Grade 3/4 toxicity rate
Disease-free survival
Time to treatment failure
1-year survival rate
2-year survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Imtiaz A. Malik, MD, Principal Investigator — Loma Linda Oncology Medical Group, Inc.
Locations (4):
- United States (4):
  - Davood Vafai, MD, Medical Offices, Incorporated, Redlands, California
  - Loma Linda Oncology Medical Group, Incorporated, Redlands, California
  - New Hope Cancer and Research Institute - Glendora, Redlands, California
  - New Hope Cancer and Research Institute - Pomona, Redlands, California